CLINICAL TRIAL: NCT03253549
Title: TecHnology Enabled Self-MAnagemenT - VIsion for Remote Automated Patient Monitoring and EmpoWerment Following Cardiac and VasculaR Surgery
Brief Title: The SMArTVIEW, CoVeRed
Acronym: SMArTVIEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Population Health Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Centres of Excellence (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMArTVIEW v1.0
Record Dates: First submitted 2017-08-10; First posted 2017-08-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Surgery (Cardiac); Surgery (Major Vascular)
Keywords: remote automated monitoring; hospital to home virtual care; cardiac surgery; major vascular surgery; self-management

STUDY DESIGN:
Intervention Model Description: Participants are randomized to SMArTVIEW or Standard Care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMArTVIEW (Experimental)
  Interventions: Device: SMArTVIEW
- Standard Care (No Intervention)

INTERVENTIONS:
Device: SMArTVIEW — Remote automated, continuous monitoring in hospital after cardiac or vascular surgery, followed by 30-day at home monitoring, daily nurse video visits and a self-management training program.
  Arms: SMArTVIEW

SUMMARY:
The SMArTVIEW program evaluates the use of remote, automated monitoring in hospital and at home, on patients undergoing cardiac and major vascular surgery, to determine the effect on the 45-day risk of a composite of hospital readmission and emergency department/urgent care centre visits (not requiring hospital admission). Half of participants will receive the SMArTVIEW intervention of increased monitoring, while the other half will receive standard care after surgery.

DETAILED DESCRIPTION:
SMArTVIEW is an eHealth-enabled service delivery program that combines remote automated monitoring, education, and self-management training. SMArTVIEW is a two-stage intervention program. Stage 1 supports seniors after cardiac or major vascular surgery in hospital on the surgical unit (post-ICU). Participants are assigned automated, cableless, vital sign monitoring devices that are worn during their entire stay on the surgical unit (blood pressure cuff, respiration pod, and oxygen saturation probe). Any signs of deterioration are sent via handheld device to the primary care nurse for early intervention.

With a view to seamless transition home, Stage 2 supports these individuals at home during the first 30 days of recovery. Participants are sent home with Bluetooth enabled monitoring equipment including a tablet, blood pressure cuff, thermometer, pulse oximeter and weight scale. From home, the tablet uploads patients' vital signs and measurements automatically and sends them, via secure cloud infrastructure, to the SMArTVIEW Nurse on the surgical ward back at the hospital. The tablet interface also prompts patients to respond to brief, easy to read, daily surveys in order to inform the nurse about their status. The tablet also supports secure daily video visits and daily interaction with the nurse for postoperative assessment and support, surgical wound photographs, as well as patient access to customized educational materials.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years;
2. Patient has undergone major cardiac or vascular surgery and has been admitted post-op to the surgical floor;
3. Anticipated length of stay (LOS) on the surgical floor is ≥ 48 hours;
4. Patient has a negative Confusion Assessment Method (CAM) test result preceding, or within 12 hours of arriving on the surgical floor and is randomized within the first 24 hours after arriving on the ward;
5. Patient is able to provide consent autonomously.

Exclusion Criteria:

1. Patient is unable to communicate with research staff, complete surveys and questionnaires, or a telephone interview;
2. Patient has an intolerance/allergy to adhesive;
3. Patient unable to complete 30 days of at-home follow up due to current or planned relocation to nursing home or rehab facility; and
4. Patients with radial graft sites

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Hospital Readmission Rate | Readmission within 45 days post discharge.
  45-day risk of a composite of hospital readmission and emergency department/urgent care centre visits (not requiring hospital admission).

SECONDARY OUTCOMES:
Composite of Major Complications associated with Undetected Hemodynamic Compromise | 45 day and 6 months post discharge
  Composite death, non-fatal myocardial infarction, non-fatal stroke, non-fatal cardiac arrest, congestive heart failure, clinically important atrial fibrillation, deep vein thrombosis or pulmonary embolism, bleeding, respiratory failure, falls, delirium, reoperation, important hypotension, acute kidney injury w/ dialysis, infection/sepsis and medication error detection and correction.
User Experience while on the SMArTVIEW Intervention compared to standard of care | 45 days and 6 months post discharge.
  Patient and clinician experience, family/caregiver experience, patient's functional status, patient activation, postoperative pain and satisfaction with care.
Econometrics | 45 days and 6 months post discharge.
  Health service utilization-related costs and patient-level of cost of recovery.
Process & Implementation | Through study completion. An average of 1 year.
  Barriers and facilitators to the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Hamilton General Hospital, Hamilton, Ontario, Canada
- Liverpool Heart & Chest Hospital, Liverpool, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided